CLINICAL TRIAL: NCT03207906
Title: A Multi-center, Randomized, Double-blind, Vehicle-controlled, Phase-2 Trial to Evaluate the Efficacy and Safety of Two Concentrations of VBP-926 Solution for the Treatment of Chemotherapy-associated Paronychia in Cancer Patients
Brief Title: A Trial to Evaluate the Efficacy and Safety of Two Concentrations of VBP-926 Solution for the Treatment of Chemotherapy-associated Paronychia in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloce BioPharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-VBP-926
Record Dates: First submitted 2017-06-28; First posted 2017-07-05 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Chemotherapy-Associated Paronychia

STUDY DESIGN:
Intervention Model Description: Once subjects have been determined to be eligible for participation in the study, they will be randomized to one of the three treatment arms. The randomization number will be generated according to the randomization schedule prepared prior to the start of the study. Participants will be assigned to receive assign treatment solution VBP-926 (either lower or higher concentration) or vehicle in 1:1:1 ratio using the IWRS system.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be done centrally by a randomization programmer/statistician who will be the only un-blinded participant. That person will not have any part in the decisions regarding patient populations and/or protocol violations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lower concentration VBP-926 (Active Comparator): VBP-926 solution applied to affected area BID
  Interventions: Drug: VBP-926
- Higher concentration VBP-926 (Active Comparator): VBP-926 solution applied to affected area BID
  Interventions: Drug: VBP-926
- Vehicle (Placebo Comparator): Vehicle solution applied to affected area BID
  Interventions: Drug: VBP-926

INTERVENTIONS:
Drug: VBP-926 — Topical VBP-926 solution

SUMMARY:
Paronychia is inflammation of the skin surrounding the nail that leads to secondary infection. Iatrogenic paronychia has been clearly associated with cancer chemotherapies. This phase-2 trial is a dose finding study and will evaluate topical VBP-926 solution against a vehicle control.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older
* Acute paronychia developing during the course of their monotherapy or combination chemotherapy
* Involvement of at least one nail with a Paronychia Severity Grading score of 1 or higher
* Eastern Cooperative Oncology Group score ≤ 2
* Life expectancy of at least 12 months as per the investigator's judgment
* Willing to provide written informed consent
* Individuals who are willing to not start any new products OTC or prescription treatments for Paronychia and discontinue any treatment the investigator feels may interfere with the evaluation of the test products
* Individuals who are already on antibiotics as prescribed by oncologist for any condition except paronychia
* Individuals who are willing to avoid using cosmetic products, creams, salves, or ointments to the treatment area(s)

Exclusion Criteria:

* Mentally incompetent or unable or not willing to give written informed consent or meet study requirements
* Without a history of a cancer diagnosis
* Without history of cancer diagnosis using chemotherapy
* Patients with paronychia requiring surgical intervention at baseline
* Patients who are already on prescribed treatment for paronychia who are not willing to discontinue this treatment and only use study drug (no washout period required)
* Neutropenia (absolute neutrophil count < 1500 cells/µL)
* Patient Human Immunodeficiency Virus (HIV) infection
* Patients with any medical condition, including alcohol or drug abuse or mental incapacity / hypersensitive to the study drug, which in judgment of the investigator will interfere with the patient's participation in the study or evaluation of study results
* Have any medical condition that, in the opinion of the investigator, may interfere with the study results or place the subject at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Downgrading of the 6-point Paronychia Severity Grading scale (adapted from CTCAE v4.0) in adult cancer patients with chemotherapy-associated paronychia | 8 weeks
  Treatment responses will be assessed by clinical grading utilizing a morphologic 6-point Paronychia Severity Grading scale (adapted from CTCAE v4.0) and will be assessed from baseline to 8 weeks for each affected nail.

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Krishnan, PhD, Study Director — JSS Research
Locations (8):
- United States (8):
  - Compassionate Cancer Care, Fountain Valley, California
  - Northwestern University Department of Dermatology, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Ohio State University, Columbus, Ohio
  - Bryn Mawr Skin & Cancer Institute, Bryn Mawr, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capriotti KD, Anadkat M, Choi J, Kaffenberger B, McLellan B, Barone S, Kukoyi O, Goldfarb S, Lacouture M. A randomized phase 2 trial of the efficacy and safety of a novel topical povidone-iodine formulation for Cancer therapy-associated Paronychia. Invest New Drugs. 2019 Dec;37(6):1247-1256. doi: 10.1007/s10637-019-00825-0. Epub 2019 Jun 26. PMID 31240513